CLINICAL TRIAL: NCT01828099
Title: A Phase III Multicenter, Randomized Study of Oral LDK378 Versus Standard Chemotherapy in Previously Untreated Adult Patients With ALK Rearranged (ALK-positive), Stage IIIB or IV, Non-squamous Non-small Cell Lung Cancer
Brief Title: LDK378 Versus Chemotherapy in Previously Untreated Patients With ALK Rearranged Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDK378A2301; 2013-000319-26 (EudraCT Number)
Record Dates: First submitted 2013-04-03; First posted 2013-04-10 (Estimated); Results first posted 2017-09-21 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; ALK; LDK378; Non-small cell lung carcinoma (NSCLC); treatment of lung cancer after first metastasis; lung cancer; lung adenocarcinoma; Non small cell lung carcinoma; Non small cell lung cancer; non-squamous non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma of Lung | interventions — ceritinib; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ceritinib (Experimental): Ceritinib administered continuously through oral dosing at a dosage of 750 mg once daily in fasted state.
  Interventions: Drug: Ceritinib
- Chemotherapy (Active Comparator): Pemetrexed plus cisplatin or carboplatin (based on Investigator's choice) for 4 cycles (Induction) followed by pemetrexed as single agent (Maintenance)
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: Ceritinib — Ceritinib was administered orally once-daily fasted at a dose of 750 mg capsules on a continuous dosing schedule.
  Other Names: LDK378
  Arms: Ceritinib
Drug: Pemetrexed — Pemetrexed was administered at a dose of 500 mg/m^2 as an intravenous (iv) infusion on Day 1 of each 21-day cycle
  Arms: Chemotherapy
Drug: Cisplatin — Cisplatin was administered by iv infusion at a dose of 75 mg/m^2 every 21 days for up to 4 cycles.
  Arms: Chemotherapy
Drug: Carboplatin — Carboplatin was administered as iv infusion (AUC 5-6) every 21 days up to 4 cycles
  Arms: Chemotherapy

SUMMARY:
To compare the efficacy and safety of ceritinib with standard first-line chemotherapy (pemetrexed plus cisplatin or carboplatin) in patients with stage IIIB (not candidates for definitive multimodality therapy) or stage IV, non-squamous non-small cell lung cancer (NSCLC) harboring a confirmed anaplastic lymphoma kinase (ALK) rearrangement, using the Ventana immunohistochemistry (IHC) test.

DETAILED DESCRIPTION:
This was an open-label, randomized, global, Phase III study that compared the efficacy and safety of ceritinib to standard first-line chemotherapy in patients with advanced (NSCLC) harboring ALK rearrangement. The confirmation of ALK rearrangement was done using the ICH test by a Novartis designated central laboratory. Prior to the study, patients had not received any previous systemic, anti-cancer therapy, including ALK inhibitors, for newly diagnosed advanced non-squamous NSCLC.

The patients were randomized in a 1:1 ratio to either receive ceritinib (750 mg once daily, fasted) or chemotherapy. The chemotherapy regimen consisted of a platinum-based doublet with pemetrexed followed by pemetrexed maintenance in patients without progressive disease after 4 cycles.

Treatment was continued until the blinded independent review committee (BIRC) confirmed disease progression based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1), occurrence of unacceptable toxicity, or meeting other discontinuation criteria. Patients in either arm were permitted to continue the assigned study treatment beyond BIRC-confirmed disease progression in case of continued clinical benefit, as determined by the Investigator.

All patients who discontinued treatment during the treatment phase for reasons other than death, lost to follow-up, pregnancy or disease progression entered the post-treatment follow-up period until disease progression, withdrawal of consent or death.

In the chemotherapy arm, patients were allowed to switch and receive ceritinib after BIRC-confirmed disease progression (extension-treatment period).

ELIGIBILITY:
Key Inclusion Criteria:

1. The patient had a histologically or cytologically confirmed diagnosis of non-squamous Non-small cell lung cancer (NSCLC) that was Anaplastic lymphoma kinase (ALK) positive as assessed by the Ventana Immunohistochemistry (IHC) test. The test was performed at Novartis designated central laboratories.
2. The patient had a newly diagnosed stage IIIB (who was not a candidate for definitive multimodality therapy) or stage IV NSCLC or relapsed locally advanced or metastatic NSCLC not previously treated with any systemic anti-cancer therapy (e.g. cytotoxic drugs, monoclonal antibody therapy, crizotinib or other ALK inhibitors, or other targeted therapies, either experimental or not), with the exception of neo-adjuvant or adjuvant therapy.
3. The patient had at least one measurable lesion as defined by RECIST 1.1.

Key Exclusion Criteria:

1. The patient had known hypersensitivity to any of the excipients of LDK378 (microcrystalline cellulose, mannitol, crospovidone, colloidal silicon dioxide, and magnesium stearate).
2. The patient had a history of severe hypersensitivity reaction to platinum-containing drugs, pemetrexed, or any known excipients of these drugs.
3. The patient had symptomatic central nervous system (CNS) metastases and was neurologically unstable or had required increasing doses of steroids within the 2 weeks prior to screening to manage CNS symptoms.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2013-07-09 (Actual); Primary Completion 2016-06-24 (Actual); Study Completion 2024-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (147):
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, La Rioja
- Australia (3):
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Auckland
- Austria (2):
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Brazil (10):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Recife, Pernambuco
  - Novartis Investigative Site, Rio de Janiero, Rio de Janeiro
  - Novartis Investigative Site, Natal, Rio Grande do Norte
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Itajaí, Santa Catarina
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São José do Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- China (10):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Guang Dong Province
  - Novartis Investigative Site, Tianjin
- Colombia (2):
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Montería
- Denmark (2):
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Odense C
- France (10):
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Toulon, Val De Marne
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Villejuif
- Germany (10):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Coswig
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Wiesbaden
- Greece (2):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Heraklion Crete
- Hungary (4):
  - Novartis Investigative Site, Zalaegerszeg, Zala County
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Veszprém
- India (11):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Madurai, Tamil Nadu
  - Novartis Investigative Site, Vellore, Tamil Nadu
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Delhi
  - Novartis Investigative Site, Mumbai
- Novartis Investigative Site, Dublin, Ireland
- Italy (15):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Napoli
- Japan (7):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Akashi, Hyōgo
  - Novartis Investigative Site, Hirakata, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Koto Ku, Tokyo
  - Novartis Investigative Site, Niigata
- Lebanon (2):
  - Novartis Investigative Site, El Achrafiyé
  - Novartis Investigative Site, Saida
- Novartis Investigative Site, Guadalajara, Jalisco, Mexico
- Netherlands (6):
  - Novartis Investigative Site, Leiden, South Holland
  - Novartis Investigative Site, Amersfroort
  - Novartis Investigative Site, Enschede
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Maastricht
  - Novartis Investigative Site, Zoetermeer
- Novartis Investigative Site, Oslo, Norway
- Poland (2):
  - Novartis Investigative Site, Szczecin
  - Novartis Investigative Site, Warsaw
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Singapore, Singapore
- South Korea (3):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Seoul
- Spain (19):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Lleida, Catalonia
  - Novartis Investigative Site, Mataró, Catalonia
  - Novartis Investigative Site, Reus, Catalonia
  - Novartis Investigative Site, Badajoz, Extremadura
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Lugo, Galicia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Sweden (4):
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- Taiwan (4):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Thailand (3):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
- United Kingdom (6):
  - Novartis Investigative Site, Exeter, Devon
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Soria JC, Tan DSW, Chiari R, Wu YL, Paz-Ares L, Wolf J, Geater SL, Orlov S, Cortinovis D, Yu CJ, Hochmair M, Cortot AB, Tsai CM, Moro-Sibilot D, Campelo RG, McCulloch T, Sen P, Dugan M, Pantano S, Branle F, Massacesi C, de Castro G Jr. First-line ceritinib versus platinum-based chemotherapy in advanced ALK-rearranged non-small-cell lung cancer (ASCEND-4): a randomised, open-label, phase 3 study. Lancet. 2017 Mar 4;389(10072):917-929. doi: 10.1016/S0140-6736(17)30123-X. Epub 2017 Jan 24. PMID 28126333
- [Derived] Lin YT, Yu CJ, Yang JC, Shih JY. Anaplastic Lymphoma Kinase (ALK) Kinase Domain Mutation Following ALK Inhibitor(s) Failure in Advanced ALK Positive Non-Small-Cell Lung Cancer: Analysis and Literature Review. Clin Lung Cancer. 2016 Sep;17(5):e77-e94. doi: 10.1016/j.cllc.2016.03.005. Epub 2016 Mar 30. PMID 27130468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled in 134 centers across 27 countries.
Pre-assignment Details: Participants had to satisfy all the inclusion criteria none of the exclusion criteria prior to randomization.
Period: Treatment Period
Arm/Group | Ceritinib | Chemotherapy
Started | 189 | 187
Treated | 189 | 175
Completed | 0 | 0
Not Completed | 189 | 187
Not completed — Adverse Event | 24 | 23
Not completed — Death | 10 | 12
Not completed — Lost to Follow-up | 2 | 1
Not completed — Non-compliance with study treatment | 1 | 0
Not completed — Physician Decision | 17 | 16
Not completed — Progressive disease | 99 | 107
Not completed — Subject/guardian decision | 22 | 26
Not completed — Study terminated by Sponsor | 13 | 1
Not completed — Protocol deviation | 1 | 0
Not completed — No longer requires treatment | 0 | 1
Period: Extension-treatment Phase
Arm/Group | Ceritinib | Chemotherapy
Started (Extension-treatment phase was for patients who crossed over from chemotherapy to ceritinib treatment.) | 0 | 102
Crossover Analysis Set (Patients who crossed over to the ceritinib arm and received at least one dose of ceritinib) | 0 | 100
Completed | 0 | 0
Not Completed | 0 | 102
Not completed — Adverse Event | 0 | 17
Not completed — Death | 0 | 11
Not completed — Physician Decision | 0 | 5
Not completed — Progressive disease | 0 | 54
Not completed — Study terminated by sponsor | 0 | 5
Not completed — Subject/guardian decision | 0 | 10

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization. According to the intent to treat principle, patients were analyzed according to the treatment and strata to which they had been assigned during the randomization procedure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceritinib | Chemotherapy | Total
Number analyzed (Participants) | 189 | 187 | 376
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (12.76) | 53.3 (12.49) | 53.9 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 114 | 216
  Male | 87 | 73 | 160
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 76 | 82 | 158
  Black | 3 | 3 | 6
  Caucasian | 104 | 98 | 202
  Native American | 3 | 2 | 5
  Other | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) by Blinded Independent Review Committee (BIRC)
Description: PFS is defined as the time from the date of randomization to the date of the first radiologically documented disease progression (as assessed by BIRC per RECIST 1.1) or death due to any cause. A patient who had not progressed or died at the date of the analysis cut-off or had received another anticancer therapy had their PFS censored at the time of the last adequate tumor evaluation before the earlier of the cut-off date or the anticancer therapy date. The distribution of PFS was estimated using the Kaplan-Meier (KM) method.
Time Frame: From the date of randomization to the date of first radiologically documented disease progression or death due to any cause, up to approximately 34 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 189 | 187
Months | 16.6 [12.6 to 27.2] | 8.1 [5.8 to 11.1]
Statistical Analysis 1: Comparison: Ceritinib vs Chemotherapy; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.42 to 0.73]

2. Secondary Outcome: Overall Survival (OS)
Description: OS defined as time from date of randomization to date of death due to any cause.
  If the patient was alive at the date of the analysis cut-off or lost to follow-up, then OS was censored at the last contact date prior to data cut-off date. The distribution of OS was estimated using the KM method.
Time Frame: From date of randomization to date of death due to any cause, up to approximately 120 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 189 | 187
Months | 62.9 [44.2 to 77.6] | 40.7 [28.5 to 54.5]

3. Secondary Outcome: Overall Response Rate (ORR) by BIRC Assessment
Description: ORR is defined as the percentage of patients with a best overall response defined as complete response (CR) or or partial response (PR) measured by BIRC per RECIST 1.1. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 34 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 189 | 187
Percentage of participants | 72.5 [65.5 to 78.7] | 26.7 [20.5 to 33.7]

4. Secondary Outcome: Overall Response Rate (ORR) by Investigator Assessment
Description: ORR is defined as the percentage of patients with a best overall response defined as complete response (CR) or or partial response (PR) measured by investigator assessment per RECIST 1.1.
  CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 120 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 189 | 187
Percentage of participants | 73.5 [66.7 to 79.7] | 33.2 [26.5 to 40.4]

5. Secondary Outcome: Duration of Response (DOR) by BIRC Assessment
Description: DOR is defined as the time from date of first documented CR or PR to date of first documented disease progression (measured by BIRC assessment per RECIST 1.1) or death due to any cause. CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  If a patient had not had an event, DOR was censored at the date of last adequate tumor assessment. Patients who had never achieved a best overall response of CR or PR were excluded from the analysis. The distribution function of DOR was estimated using the KM method.
Time Frame: From first documented response to first documented disease progression or death, assessed up to approximately 34 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization. Patients with confirmed CR or PR by BIRC assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 137 | 50
Months | 23.9 [16.6 to NA] — NA: not estimable due to an insufficient number of participants with events. | 11.1 [7.8 to 16.4]

6. Secondary Outcome: Duration of Response (DOR) by Investigator Assessment
Description: DOR is defined as the time from date of first documented CR or PR to date of first documented disease progression (measured by investigator assessment per RECIST 1.1) or death due to any cause.
  CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  If a patient had not had an event, DOR was censored at the date of last adequate tumor assessment. Patients who had never achieved a best overall response of CR or PR were excluded from the analysis. The distribution function of DOR was estimated using the KM method.
Time Frame: From first documented response to first documented disease progression or death, assessed up to approximately 120 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization. Patients with confirmed CR or PR by investigator assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 139 | 62
Months | 22.6 [17.7 to 26.2] | 9.8 [6.1 to 16.9]

7. Secondary Outcome: Disease Control Rate (DCR) by BIRC Assessment
Description: DCR is defined as the percentage of patients with best overall response of CR, PR, or stable disease (SD) measured by BIRC assessment per RECIST 1.1.
  CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Up to approximately 34 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 189 | 187
Percentage of participants | 84.7 [78.7 to 89.5] | 73.8 [66.9 to 79.9]

8. Secondary Outcome: Disease Control Rate (DCR) by Investigator Assessment
Description: DCR is defined as the percentage of patients with best overall response of CR, PR, or stable disease (SD) measured by investigator assessment per RECIST 1.1.
  CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Up to approximately 120 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 189 | 187
Percentage of participants | 89.4 [84.1 to 93.4] | 75.9 [69.2 to 81.9]

9. Secondary Outcome: Time to Response (TTR) by BIRC Assessment
Description: TTR is defined as the time from date of randomization to date of first documented response (CR or PR) measured by BIRC assessment per RECIST 1.1.
  CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  Patients who had not achieved a confirmed CR or PR were censored at the last adequate tumor assessment date when they had not had a PFS event or at maximum follow-up when they had had a PFS event.
Time Frame: From randomization to date of first documented response, up to approximately 34 months
Population: as for outcome 5
Measure: Median (Full Range); unit: Weeks
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 137 | 50
Weeks | 6.14 [5.1 to 61.7] | 13.36 [5.1 to 90.1]

10. Secondary Outcome: Time to Response (TTR) by Investigator Assessment
Description: TTR is defined as the time from date of randomization to date of first documented response (CR or PR) measured by investigator assessment per RECIST 1.1.
  CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  Patients who had not achieved a confirmed CR or PR were censored at the last adequate tumor assessment date when they had not had a PFS event or at maximum follow-up when they had had a PFS event
Time Frame: From randomization to date of first documented response, up to approximately 120 months
Population: as for outcome 6
Measure: Median (Full Range); unit: Weeks
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 139 | 62
Weeks | 6.29 [5.1 to 71.9] | 12.71 [4.7 to 461.6]

11. Secondary Outcome: PFS by Investigator Assessment
Description: PFS is defined as the time from the date of randomization to the date of the first radiologically documented disease progression (as assessed by investigator assessment per RECIST 1.1) or death due to any cause.
  A patient who had not progressed or died at the date of the analysis cut-off or had received another anticancer therapy had their PFS censored at the time of the last adequate tumor evaluation before the earlier of the cut-off date or the anticancer therapy date. The distribution of PFS was estimated using the KM method.
Time Frame: From the date of randomization to the date of first radiologically documented disease progression or death due to any cause, up to approximately 120 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 189 | 187
Months | 16.8 [13.5 to 22.8] | 7.2 [5.8 to 9.7]

12. Secondary Outcome: Overall Intracranial Response Rate (OIRR)
Description: OIRR is defined as the ORR based on lesions in brain (target, non-target lesions and new lesions, if applicable) and calculated as the percentage of patients with a best overall confirmed response of CR or PR in the brain per modified RECIST 1.1 as assessed by BIRC neuroradiologist.
  CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 34 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization. Patients with measurable brain disease and who had a baseline and at least one post-baseline scan
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 22 | 22
Percentage of participants | 72.7 [49.8 to 89.3] | 27.3 [10.7 to 50.2]

13. Secondary Outcome: Intracranial Disease Control Rate (IDCR)
Description: IDCR is defined as the DCR based on lesions in brain (target, non-target lesions and new lesions, if applicable) and calculated as the percentage of patients with a best overall response of CR or PR or SD (or non-CR/nonPD) in the brain per modified RECIST 1.1 as assessed by BIRC neuro-radiologist.
  CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease
Time Frame: Up to approximately 34 months
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 22 | 22
Percentage of participants | 86.4 [65.1 to 97.1] | 90.9 [70.8 to 98.9]

14. Secondary Outcome: Duration of Intracranial Response (DOIR)
Description: DOIR is defined as the DOR based on lesions in brain (target, non-target lesions and new lesions, if applicable) and calculated from the time of first documented response of CR or PR to the date of the first documented disease progression in the brain or death due to any cause per modified RECIST 1.1 as assessed by BIRC neuro-radiologist.
  CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From first documented response to first documented disease progression in the brain or death, assessed up to approximately 34 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization. Patients with measurable brain disease and who had a baseline and at least one post-baseline scan, and a confirmed intracranial CR or PR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 16 | 6
Months | 16.6 [8.1 to NA] — NA: not estimable due to an insufficient number of participants with events. | NA [1.5 to NA] — NA: not estimable due to an insufficient number of participants with events.

15. Secondary Outcome: Time to Definitive 10 Point Deterioration in the Composite Endpoint of Pain, Cough or Dyspnea in the European Organization for Research and Treatment of Cancer Quality of Life (EORTC QLQ)- Lung Cancer (LC) 13 Questionnaire
Description: The EORTC QLQ-LC13 complemented the QLQ-C30 and measured disease symptoms and treatment-related adverse effects. The lung cancer module incorporated one multi-item scale to assess dyspnea and 9 single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. All of the domain scores ranged from 0 to 100. A high score indicated a high level of symptoms.
  Time to definitive symptom deterioration for the composite endpoint was defined as the time from the date of randomization to the earliest date when the patient's score showed a 10 point or higher increase from baseline in any of the symptoms (pain, cough or dyspnea) as per EORTC QLQ-LC13 (with no later change below this threshold i.e., <10 points was observed or if this increase was observed at the last assessment for the patient) or death due to any cause.
Time Frame: Screening, treatment phase (Cycles 2, 3 then every 2nd cycle until Month 33; after Month 33, every 9 or 12 weeks, end of treatment); follow-up phase (Every 6 weeks until Month 33; after Month 33 every 9 or 12 weeks) up to approximately 120 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 189 | 187
Months | 76.0 [42.2 to NA] — NA: not estimable due to an insufficient number of participants with events. | 14.9 [11.1 to 27.7]

16. Secondary Outcome: Time to Definitive Deterioration in the Composite Endpoint of Pain, Cough or Dyspnea in the Lung Cancer Symptom Scale (LCSS)
Description: The LCSS patient scale used a 24-hour recall period and contained nine items: six measuring major symptoms for lung cancer (appetite loss, fatigue, cough, dyspnea, hemoptysis, pain), and three summary items related to total symptom distress, normal activity status, and overall quality of life. The LCSS used a 100mm visual analog scale (VAS) to measure the intensity of patient responses, with zero corresponding to the lowest rating (best status) and 100 representing the highest rating (worst status).
  Time to definitive deterioration for the composite endpoint was defined as the time from the date of randomization to the earliest date when the patient's score showed a 10 point or higher increase from baseline in any of the LCSS scores related to pain in the chest, cough, or dyspnea (with no later change below this threshold i.e., <10 points was observed or if this increase was observed at the last assessment for the patient) or death due to any cause.
Time Frame: as for outcome 15
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 189 | 187
Months | 104.0 [76.0 to NA] — NA: not estimable due to an insufficient number of participants with events. | 36.1 [18.4 to 100.8]

17. Secondary Outcome: Least Squares Mean Scores on the EORTC-QLQ C30
Description: The EORTC QLQ-C30 contained 30 items and was of both multi-item scales and single-item measures, including 5 functional scales (physical, role, emotional, cognitive, and social functioning), 3 symptom scales (fatigue, nausea/vomiting, and pain), 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties), and a global health status (GHS)/quality of life (QoL) scale. Items were assessed on a 4- or 7-level Likert scale, ranging from 1="very poor" to 7= "excellent" for GHS items and 1= "not at all" to 4= "very much" for all other items. The scores of the scales were averaged from the scores of the component items, transformed, and analyzed on a 0 - 100 scale. A high score represented a higher response level. The scores were analyzed using repeated measurement model for longitudinal data, including terms for visit, treatment, treatment by time interaction, strata and baseline score. Overall mean and standard error were obtained
Time Frame: as for outcome 15
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization. Participants with a baseline assessment for at least one of the scales/single items
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 182 | 161
Score on a scale
  Global Health Status/QoL: number analyzed (Participants) | 181 | 161
  Global Health Status/QoL | 69.4 (0.71) | 63.7 (0.98)
  Physical Functioning | 83.5 (0.78) | 77.6 (1.07)
  Emotional Functioning: number analyzed (Participants) | 181 | 161
  Emotional Functioning | 82.3 (0.70) | 76.6 (0.97)
  Social Functioning: number analyzed (Participants) | 181 | 161
  Social Functioning | 79.0 (1.01) | 75.4 (1.38)
  Cognitive Functioning: number analyzed (Participants) | 181 | 161
  Cognitive Functioning | 86.7 (0.68) | 84.0 (0.94)
  Role Functioning | 79.5 (1.03) | 71.3 (1.44)
  Fatigue | 25.9 (0.84) | 31.4 (1.17)
  Nausea and Vomiting | 11.8 (0.58) | 11.6 (0.82)
  Pain: number analyzed (Participants) | 181 | 161
  Pain | 14.7 (0.75) | 16.9 (1.05)
  Dyspnea | 15.0 (0.75) | 22.1 (1.05)
  Insomnia | 14.8 (0.78) | 21.1 (1.09)
  Appetite Loss | 15.9 (0.82) | 19.3 (1.15)
  Constipation | 8.1 (0.60) | 13.0 (0.84)
  Diarrhea: number analyzed (Participants) | 181 | 161
  Diarrhea | 25.7 (0.80) | 4.6 (1.12)
  Financial Difficulties: number analyzed (Participants) | 181 | 160
  Financial Difficulties | 19.9 (1.19) | 23.8 (1.63)

18. Secondary Outcome: Least Squares Mean Scores on the EORTC QLQ- LC13
Description: The EORTC QLQ-LC13 was used in conjunction with the EORTC QLQ-C30 and provided information on an additional 13 items specifically related to lung cancer. The lung cancer module incorporated one multi-item scale to assess dyspnea, and 9 single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. Items were scored on a 4-point Likert scale ranging from 1="not at all" to 4="very much". For the multi-item scale, the scores were averaged from the scores of the component items, transformed, and then analyzed on a 0 - 100 scale. For the single item scale, raw scores were transformed and analyzed on a 0-100 scale. A high score indicated a high level of symptoms The scores were analyzed using repeated measurement model for longitudinal data, including terms for visit, treatment, treatment by time interaction, strata and baseline score. Overall mean and standard error were obtained.
Time Frame: as for outcome 15
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization. Participants with a baseline assessment for at least one of the domain scores
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 181 | 159
Score on a scale
  Dyspnoea: number analyzed (Participants) | 181 | 158
  Dyspnoea | 16.2 (0.74) | 23.3 (1.02)
  Pain in chest | 9.4 (0.59) | 11.8 (0.82)
  Pain in Arm or Shoulder: number analyzed (Participants) | 181 | 157
  Pain in Arm or Shoulder | 10.6 (0.69) | 12.3 (0.97)
  Pain in Other Parts: number analyzed (Participants) | 180 | 157
  Pain in Other Parts | 12.5 (0.71) | 15.0 (1.01)
  Coughing | 14.7 (0.63) | 23.0 (0.88)
  Sore Mouth | 3.0 (0.35) | 6.8 (0.49)
  Dysphagia | 4.1 (0.37) | 5.5 (0.52)
  Peripheral Neuropathy | 9.7 (0.69) | 16.0 (0.96)
  Alopecia | 6.8 (0.70) | 13.3 (0.95)
  Haemoptysis | 0.7 (0.18) | 1.5 (0.25)

19. Secondary Outcome: Least Squares Mean Scores on the Lung Cancer Symptom Scale (LCSS)
Description: The LCSS consisted of 9 individual items; 6 measured lung cancer symptoms (appetite, fatigue, cough, dyspnea, hemoptysis, and pain); the remaining 3 items measured general lung cancer symptom distress, interference with daily activities and overall QoL. Each item was scored on a 100-millimeter Visual Analogue Scale (VAS), with scores ranging from 0 to 100 (0 = best outcome).
  Total score was calculated as the average of the aggregate score of all 9 items. Scores ranged from 0 to 100, with higher total scores indicating a greater overall impact of symptoms on the patient's QoL. The Symptom Burden Index (SBI) was calculated as the average of the six symptom items. It also ranged from 0 to 100, with higher scores indicating greater symptom burden.
  Scores were analyzed using repeated measurement model for longitudinal data, including terms for visit, treatment, treatment by time interaction, strata and baseline score. Overall mean and standard error were obtained.
Time Frame: as for outcome 15
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 183 | 161
Score on a Scale
  Appetite Loss | 20.9 (1.35) | 25.1 (1.58)
  Fatigue | 27.4 (1.50) | 33.9 (1.74)
  Cough | 8.0 (0.87) | 15.1 (1.02)
  Shortness of Breath | 18.8 (1.40) | 25.5 (1.62)
  Hemoptysis: number analyzed (Participants) | 183 | 160
  Hemoptysis | 0.7 (0.37) | 1.9 (0.44)
  Pain | 11.6 (1.16) | 14.9 (1.35)
  Total Symptom Distress: number analyzed (Participants) | 182 | 161
  Total Symptom Distress | 20.5 (1.75) | 29.3 (2.02)
  Normal Activity Status | 23.6 (1.59) | 33.5 (1.84)
  Overall Quality of Life: number analyzed (Participants) | 182 | 161
  Overall Quality of Life | 27.4 (1.56) | 35.3 (1.75)
  Symptom Burden Index: number analyzed (Participants) | 183 | 160
  Symptom Burden Index | 14.7 (0.91) | 19.4 (1.05)
  Total Score: number analyzed (Participants) | 181 | 160
  Total Score | 19.1 (1.18) | 24.7 (1.31)

20. Secondary Outcome: Least Squares Mean Scores on the EQ-5D-5L Index
Description: The EQ-5D-5L descriptive system provides a profile of the participant's health state in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each of these dimensions, the participant self-assigned a score: from 1 (no problems) to 5 (extreme problems). The 5 digit health states obtained for each dimension was converted into a single mean index value based on the EQ-5D crosswalk value set for the UK using the time trade-off method. This index ranges from -0.594 (worst health) to 1.0 (best health).
  The scores were analyzed using repeated measurement model for longitudinal data, including terms for visit, treatment, treatment by time interaction, strata and baseline score. Overall mean and standard error were obtained.
Time Frame: as for outcome 15
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization. Participants with a baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 180 | 159
Score on a Scale | 0.80 (0.01) | 0.75 (0.01)

21. Secondary Outcome: Least Squares Mean Scores on the EQ-5D-5L Visual Analogue Score (VAS)
Description: The EQ-5D-5L questionnaire is a standardized measure of health status. The EQ-5D-5L descriptive system comprises of the 5 following dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Along with the five dimensions of health, the EQ-5D-5L includes a VAS where respondents rate their overall health status on a scale from 0 to 100, where 0 represents the worst possible health state and 100 represents the best possible health state. A positive change from baseline indicates improvement.
  The scores were analyzed using repeated measurement model for longitudinal data, including terms for visit, treatment, treatment by time interaction, strata and baseline score. Overall mean and standard error were obtained.
Time Frame: as for outcome 15
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 180 | 156
Score on a Scale | 77.2 (0.65) | 74.1 (0.90)

22. Secondary Outcome: Cmax of LDK378
Description: The observed maximum plasma concentration following administration
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 at pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose. Cycle=21 days
Population: The Pharmacokinetic Analysis Set (PAS) consisted of all patients who received at least one (full or partial) dose of LDK378 and provided at least one evaluable pharmacokinetic (PK) blood sample. Only the subset of participants with extensive PK collection were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng) / mililiter (ml)
Arm/Group | Ceritinib
Number analyzed (Participants) | 7
nanogram (ng) / mililiter (ml)
  Cycle 1 Day 1 | 162 (106.9)
  Cycle 2 Day 1: number analyzed (Participants) | 6
  Cycle 2 Day 1 | 794 (39.2)

23. Secondary Outcome: Tmax of LDK378
Description: The time to reach peak or maximum concentration (Tmax) was assessed. Actual recorded sampling times were considered for the calculations
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 at pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose. Cycle=21 days
Population: The Pharmacokinetic Analysis Set (PAS) consisted of all patients who received at least one (full or partial) dose of LDK378 and provided at least one evaluable PK blood sample. Only the subset of participants with extensive PK collection were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Ceritinib
Number analyzed (Participants) | 7
hours
  Cycle 1 Day 1 | 6.00 [4.00 to 8.00]
  Cycle 2 Day 1: number analyzed (Participants) | 6
  Cycle 2 Day 1 | 6.00 [6.00 to 24.00]

24. Secondary Outcome: Tlast of LDK378
Description: The time to last quantifiable concentration. Actual recorded sampling times were considered for the calculations
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 at pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose. Cycle=21 days
Population: as for outcome 23
Measure: Median (Full Range); unit: Hours
Arm/Group | Ceritinib
Number analyzed (Participants) | 7
Hours
  Cycle 1 Day 1 | 24.0 [23.7 to 24.2]
  Cycle 2 Day 1: number analyzed (Participants) | 6
  Cycle 2 Day 1 | 24.0 [23.8 to 24.3]

25. Secondary Outcome: AUC0-24 of LDK378
Description: The area under the plasma concentration-time curve calculated from time zero to 24 hours
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 at pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose. Cycle=21 days
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Ceritinib
Number analyzed (Participants) | 7
hours*ng/mL
  Cycle 1 Day 1 | 2540 (113.1)
  Cycle 2 Day 1: number analyzed (Participants) | 6
  Cycle 2 Day 1 | 16600 (44.0)

26. Post Hoc Outcome: All Collected Deaths
Description: Pre-treatment: From randomization to start of treatment. On-Treatment: From start of treatment to 30 days post-treatment or start of crossover treatment.
  Extension-treatment: From start of crossover treatment to 30 days post-crossover treatment.
  Post-treatment: From 31 days after last dose of treatment to the end of study.
Time Frame: Pre-treatment: up to 28 days; On-Treatment: up to approx. 120 months; Extension-treatment: up to approx. 108 months; Post-treatment: up to approx. 120 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
  For the Chemotherapy/Ceritinib group, the analysis included patients randomized to the chemotherapy arm who crossed over and received at least one dose of ceritinib
Measure: Count of Participants; unit: Participants
Groups:
- Chemotherapy to Ceritinib: Patients randomized to chemotherapy who crossed over to ceritinib at the extension-treatment period
Arm/Group | Ceritinib | Chemotherapy | Chemotherapy to Ceritinib
Number analyzed (Participants) | 189 | 187 | 100
Participants
  Pre-treatment: number analyzed (Participants) | 189 | 187 | 0
  Pre-treatment | 0 | 3 | 0
  On-Treatment: number analyzed (Participants) | 189 | 175 | 100
  On-Treatment | 15 | 7 | 15
  Post-treatment: number analyzed (Participants) | 149 | 60 | 83
  Post-treatment | 98 | 38 | 56
  All deaths | 113 | 48 | 71

ADVERSE EVENTS:
Time Frame: All-cause mortality: from randomization up to approx. 120 months, including post-treatment survival follow-up period. Serious and Other Adverse Events (AEs): from first dose of study treatment until 30 days after last dose (or start of crossover treatment), up to approx. 120 months. For participants who crossed over, AEs were also collected from start of crossover treatment to 30 days post-crossover treatment (extension-treatment period), up to approx. 108 months.
Description: All-cause mortality: reported for all randomized participants regardless of whether the assigned study treatment was received. Deaths in post-treatment survival follow-up period (more than 30 days after last dose) are reported separately and are not considered AEs.
  Serious and Other AEs: reported for all randomized participants who received at least one dose of study treatment
Groups:
- Ceritinib: All-cause mortality from randomization until 30 days after last dose. Adverse Events from first dose until 30 days after last dose.
- Chemotherapy: All-cause mortality from randomization until 30 days after last dose or start of crossover treatment. Adverse Events from first dose until 30 days after last dose or start of crossover treatment.
- Chemotherapy to Ceritinib (Extension-treatment): All-cause mortality and Adverse Events from start of crossover treatment to 30 days post-crossover treatment
- Ceritinib (Post-treatment Follow-up); Chemotherapy (Post-treatment Follow-up): Deaths collected in the post- treatment survival follow-up period (starting from day 31 after last dose). No AEs were collected during this period
- Chemotherapy to Ceritinib (Post-treatment Follow-up): Deaths collected in the post- treatment survival follow-up period (starting from day 31 after last dose of crossover treatment). No AEs were collected during this period
Arm/Group | Ceritinib | Chemotherapy | Chemotherapy to Ceritinib (Extension-treatment) | Ceritinib (Post-treatment Follow-up) | Chemotherapy (Post-treatment Follow-up) | Chemotherapy to Ceritinib (Post-treatment Follow-up)
All-Cause Mortality (participants affected / at risk) | 15/189 | 10/187 | 15/100 | 98/149 | 38/60 | 56/83
Serious Adverse Events (participants affected / at risk) | 93/189 | 64/175 | 47/100 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 186/189 | 166/175 | 99/100 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ceritinib (N=189) | Chemotherapy (N=175) | Chemotherapy to Ceritinib (Extension-treatment) (N=100) | Ceritinib (Post-treatment Follow-up) (N=0) | Chemotherapy (Post-treatment Follow-up) (N=0) | Chemotherapy to Ceritinib (Post-treatment Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 1 | NA | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | NA | NA | NA
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | NA | NA | NA
Atrial fibrillation (Cardiac disorders) | 2 | 2 | 0 | NA | NA | NA
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | NA | NA | NA
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | NA | NA | NA
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 1 | NA | NA | NA
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | NA | NA | NA
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | NA | NA | NA
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Nodal rhythm (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Palpitations (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Pericardial effusion (Cardiac disorders) | 4 | 2 | 2 | NA | NA | NA
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 0 | NA | NA | NA
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 1 | 0 | NA | NA | NA
Blindness (Eye disorders) | 0 | 1 | 0 | NA | NA | NA
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 1 | NA | NA | NA
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 1 | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 6 | 5 | 0 | NA | NA | NA
Oesophageal spasm (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 7 | 6 | 2 | NA | NA | NA
Asthenia (General disorders) | 1 | 0 | 0 | NA | NA | NA
Chest discomfort (General disorders) | 0 | 1 | 0 | NA | NA | NA
Death (General disorders) | 1 | 0 | 0 | NA | NA | NA
Fatigue (General disorders) | 2 | 3 | 3 | NA | NA | NA
General physical health deterioration (General disorders) | 2 | 0 | 2 | NA | NA | NA
Malaise (General disorders) | 2 | 1 | 1 | NA | NA | NA
Non-cardiac chest pain (General disorders) | 1 | 0 | 2 | NA | NA | NA
Pyrexia (General disorders) | 2 | 5 | 3 | NA | NA | NA
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0 | 0 | NA | NA | NA
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | NA | NA | NA
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | NA | NA | NA
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1 | NA | NA | NA
Liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Acute hepatitis B (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Appendicitis (Infections and infestations) | 1 | 1 | 0 | NA | NA | NA
Arthritis infective (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Brain abscess (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Bronchitis (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
COVID-19 (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Cellulitis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Diarrhoea infectious (Infections and infestations) | 1 | 1 | 1 | NA | NA | NA
Erysipelas (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Eye abscess (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Febrile infection (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Gastroenteritis (Infections and infestations) | 1 | 1 | 1 | NA | NA | NA
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Helicobacter gastritis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Influenza (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Localised infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | NA | NA | NA
Lung abscess (Infections and infestations) | 2 | 0 | 0 | NA | NA | NA
Lymphangitis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Mastoiditis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Meningitis bacterial (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Otitis media acute (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Peritonitis (Infections and infestations) | 0 | 1 | 1 | NA | NA | NA
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Pneumonia (Infections and infestations) | 13 | 9 | 8 | NA | NA | NA
Pneumonia aspiration (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Pyomyositis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | NA | NA | NA
Salmonella sepsis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Sepsis (Infections and infestations) | 0 | 2 | 1 | NA | NA | NA
Septic shock (Infections and infestations) | 0 | 2 | 1 | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | NA | NA | NA
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | NA | NA | NA
Viral infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | NA | NA | NA
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Post procedural oedema (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Radiation necrosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 3 | 0 | 3 | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 4 | 0 | 3 | NA | NA | NA
Blood creatinine increased (Investigations) | 3 | 0 | 2 | NA | NA | NA
Blood potassium decreased (Investigations) | 0 | 1 | 0 | NA | NA | NA
C-reactive protein increased (Investigations) | 1 | 0 | 0 | NA | NA | NA
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 1 | NA | NA | NA
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 0 | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | NA | NA | NA
Liver function test abnormal (Investigations) | 0 | 0 | 2 | NA | NA | NA
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | NA | NA | NA
Transaminases increased (Investigations) | 0 | 1 | 0 | NA | NA | NA
Weight decreased (Investigations) | 1 | 0 | 0 | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 0 | NA | NA | NA
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 1 | 2 | NA | NA | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | NA | NA | NA
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | NA | NA | NA
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | NA | NA | NA
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | NA | NA | NA
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | NA | NA | NA
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0 | 0 | NA | NA | NA
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | NA | NA | NA
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | NA | NA | NA
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Dizziness (Nervous system disorders) | 2 | 0 | 0 | NA | NA | NA
Epilepsy (Nervous system disorders) | 3 | 0 | 0 | NA | NA | NA
Headache (Nervous system disorders) | 1 | 1 | 0 | NA | NA | NA
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Paraesthesia (Nervous system disorders) | 2 | 0 | 0 | NA | NA | NA
Paraparesis (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Sciatica (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Seizure (Nervous system disorders) | 0 | 1 | 4 | NA | NA | NA
Somnolence (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Spinal cord compression (Nervous system disorders) | 0 | 1 | 1 | NA | NA | NA
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | NA | NA | NA
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | NA | NA | NA
Depression (Psychiatric disorders) | 1 | 0 | 0 | NA | NA | NA
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | NA | NA | NA
Gastrointestinal somatic symptom disorder (Psychiatric disorders) | 0 | 1 | 0 | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 5 | NA | NA | NA
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0 | NA | NA | NA
Hydronephrosis (Renal and urinary disorders) | 2 | 0 | 0 | NA | NA | NA
Renal failure (Renal and urinary disorders) | 2 | 0 | 2 | NA | NA | NA
Renal tubular disorder (Renal and urinary disorders) | 0 | 1 | 0 | NA | NA | NA
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | NA | NA | NA
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | NA | NA | NA
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 8 | 3 | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | NA | NA | NA
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 2 | NA | NA | NA
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | NA | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | NA | NA | NA
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 1 | NA | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2 | NA | NA | NA
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Circulatory collapse (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | NA | NA | NA
Embolism (Vascular disorders) | 0 | 1 | 0 | NA | NA | NA
Hypotension (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0 | NA | NA | NA
Superior vena cava syndrome (Vascular disorders) | 0 | 2 | 0 | NA | NA | NA
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ceritinib (N=189) | Chemotherapy (N=175) | Chemotherapy to Ceritinib (Extension-treatment) (N=100) | Ceritinib (Post-treatment Follow-up) (N=0) | Chemotherapy (Post-treatment Follow-up) (N=0) | Chemotherapy to Ceritinib (Post-treatment Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 34 | 63 | 21 | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 7 | 17 | 6 | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 13 | 42 | 10 | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 17 | 4 | NA | NA | NA
Tinnitus (Ear and labyrinth disorders) | 4 | 16 | 4 | NA | NA | NA
Lacrimation increased (Eye disorders) | 2 | 10 | 1 | NA | NA | NA
Abdominal distension (Gastrointestinal disorders) | 17 | 4 | 3 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 50 | 14 | 17 | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 49 | 11 | 12 | NA | NA | NA
Constipation (Gastrointestinal disorders) | 39 | 39 | 17 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 160 | 17 | 76 | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 18 | 11 | 7 | NA | NA | NA
Haemorrhoids (Gastrointestinal disorders) | 7 | 9 | 0 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 130 | 99 | 49 | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 16 | 19 | 6 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 127 | 59 | 54 | NA | NA | NA
Asthenia (General disorders) | 36 | 38 | 14 | NA | NA | NA
Face oedema (General disorders) | 3 | 10 | 1 | NA | NA | NA
Fatigue (General disorders) | 62 | 53 | 27 | NA | NA | NA
Influenza like illness (General disorders) | 12 | 4 | 4 | NA | NA | NA
Non-cardiac chest pain (General disorders) | 41 | 18 | 8 | NA | NA | NA
Oedema peripheral (General disorders) | 15 | 32 | 11 | NA | NA | NA
Pyrexia (General disorders) | 43 | 22 | 14 | NA | NA | NA
Bronchitis (Infections and infestations) | 11 | 4 | 2 | NA | NA | NA
Influenza (Infections and infestations) | 18 | 8 | 4 | NA | NA | NA
Nasopharyngitis (Infections and infestations) | 22 | 12 | 7 | NA | NA | NA
Pneumonia (Infections and infestations) | 15 | 6 | 7 | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 28 | 21 | 9 | NA | NA | NA
Urinary tract infection (Infections and infestations) | 11 | 8 | 6 | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 121 | 40 | 53 | NA | NA | NA
Amylase increased (Investigations) | 28 | 12 | 16 | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 103 | 34 | 48 | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 58 | 11 | 25 | NA | NA | NA
Blood bilirubin increased (Investigations) | 14 | 1 | 1 | NA | NA | NA
Blood creatinine increased (Investigations) | 53 | 20 | 43 | NA | NA | NA
Creatinine renal clearance decreased (Investigations) | 14 | 6 | 10 | NA | NA | NA
Electrocardiogram QT prolonged (Investigations) | 27 | 2 | 7 | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 70 | 19 | 30 | NA | NA | NA
Haemoglobin decreased (Investigations) | 7 | 13 | 5 | NA | NA | NA
Lipase increased (Investigations) | 17 | 2 | 5 | NA | NA | NA
Neutrophil count decreased (Investigations) | 6 | 30 | 3 | NA | NA | NA
Platelet count decreased (Investigations) | 6 | 11 | 0 | NA | NA | NA
Weight decreased (Investigations) | 51 | 26 | 19 | NA | NA | NA
White blood cell count decreased (Investigations) | 11 | 34 | 3 | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 67 | 59 | 21 | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 24 | 14 | 12 | NA | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 4 | 7 | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 8 | 10 | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 13 | 11 | 6 | NA | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 11 | 0 | 3 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 46 | 28 | 14 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 47 | 30 | 14 | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 6 | NA | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 | 2 | 1 | NA | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11 | 1 | 6 | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 15 | 5 | 4 | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 9 | 2 | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 16 | 3 | 3 | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 37 | 15 | 6 | NA | NA | NA
Dizziness (Nervous system disorders) | 35 | 17 | 8 | NA | NA | NA
Dysgeusia (Nervous system disorders) | 16 | 11 | 4 | NA | NA | NA
Headache (Nervous system disorders) | 46 | 23 | 17 | NA | NA | NA
Paraesthesia (Nervous system disorders) | 13 | 11 | 2 | NA | NA | NA
Anxiety (Psychiatric disorders) | 10 | 5 | 2 | NA | NA | NA
Insomnia (Psychiatric disorders) | 22 | 20 | 11 | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 58 | 33 | 20 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 35 | 30 | 17 | NA | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 14 | 13 | 3 | NA | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 8 | 4 | NA | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 | 8 | 6 | NA | NA | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 12 | 5 | 3 | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 13 | 16 | 2 | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 7 | 6 | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 25 | 10 | 7 | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 36 | 15 | 19 | NA | NA | NA
Hypertension (Vascular disorders) | 15 | 14 | 8 | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.